CLINICAL TRIAL: NCT05377112
Title: A Double-Blind, Randomized, Placebo-controlled Study to Assess the Safety, Tolerability, and Pharmacodynamics of SYNB8802v1 in Subjects With History of Gastric Bypass Surgery or Short-bowel Syndrome
Brief Title: Safety, Tolerability, and Pharmacodynamics of SYNB8802v1 in Subjects With History of Gastric Bypass Surgery or Short-bowel Syndrome
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Synlogic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SYNB8802-CP-002
Record Dates: First submitted 2022-04-15; First posted 2022-05-17 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Enteric Hyperoxaluria

STUDY DESIGN:
Intervention Model Description: Placebo control (3:2 [active: placebo]) is included for a better understanding of the safety and tolerability of SYNB8802v1.
Who Masked: Participant, Investigator
Masking Description: double-blind (sponsor-open),
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SYNB8802v1 (Experimental): Dose ramp to 1 × 1011 QD and then dose ramp to 3 × 1011 TID SYNB8802v1 live cells
  Interventions: Drug: SYNB8802v1
- Placebo (Placebo Comparator): Placebo will be administered during the dose ramp such that all subjects receive IMP dosing TID
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: SYNB8802v1 — SYNB8802v1 is an orally administered, non-systemically absorbed live biotherapeutic developed for the treatment of EH. The strain converts oxalate to formate and CO2, two naturally occurring GI metabolites.
  SYNB8802 was developed by engineering a pathway for oxalate degradation in a probiotic strain of Escherichia coli Nissle 1917 (EcN). It is intended to act within the GI tract to reduce the oxalate levels in patients with EH by converting oxalate to formate and CO2, two naturally occurring GI metabolites.
  Arms: SYNB8802v1
Other: Placebo — placebo powder will be aliquoted into high density polyethylene (HDPE) bottles and diluted in the same formulation buffer as SYNB8802v1 lyophilized powder. The placebo consists of corn starch and dyes to color match the placebo to the SYNB8802v1 powder for oral suspension
  Arms: Placebo

SUMMARY:
Study SYNB8802-CP-002 is designed to assess safety, tolerability, and oxalate lowering, in subjects with a history of gastric bypass surgery or short-bowel syndrome. In addition, this study will explore other PD effects relative to baseline as well as predictors of efficacy and tolerability.

DETAILED DESCRIPTION:
This is a double-blind (sponsor-open), randomized (3:2), placebo-controlled, inpatient study evaluating the safety and tolerability of SYNB8802v1 in subjects with a history of gastric bypass surgery or short-bowel syndrome. An interim analysis of results by an unblinded statistician will be performed after 10 subjects.

The study includes the following periods:

* Screening period (27 days)
* Diet run in (3 days)
* Dosing Period (12 days)
* Safety follow-up (28 days)

The maximum duration of the inpatient stay will be 17 days (Day -4 to Day 13). Subjects will report to the clinical research unit (CRU) on Day -4 and will complete a 3-day diet run-in period (Days -3 to -1) during which they will consume an AOLC diet (refer to Diet Manual for details). Dietary oxalate and calcium will be distributed across 3 meals per day, and subjects will maintain this diet until the end of the dosing period. A proton pump inhibitor (PPI, esomeprazole) will be administered once daily (QD), 60-90 minutes before breakfast, from the start of the diet run-in period (Day -3) until the end of the dosing period (Day 12).

On Day 1, subjects will be randomly assigned to treatment with SYNB8802v1 or placebo (collectively referred to as investigational medicinal product [IMP]). The dosing period consists of 12 days following a dose escalation plan from 1 × 1011 live cells QD to 3 × 1011 live cells TID; the dosing period for each dose level includes a 2-day dose ramp and a 3-day steady-state period. During the dose ramp, placebo will be administered such that all subjects receive IMP dosing TID. On the morning of the first day of the run-in period (Day -3), a forced void urine sample will be collected to completely empty the bladder before the first placebo dose administration. A 24-hour urine collection will then be started and will continue throughout the in-patient period. In addition, daily 24-hour fecal samples will be collected. Subjects will be released from the CRU upon the completion of safety assessments on Day 13 (the day after the last dose of IMP). Safety follow-up visits (calls) will occur every 7 (±2) days until 28 (±2) days after the last dose of IMP.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 to ≤ 74 years.
* Able and willing to voluntarily complete the informed consent process.
* Available for, and agree to, all study procedures, including fixed diet, feces, urine, and blood
* collection, follow-up visits, and compliance with all study procedures.
* History of gastric bypass surgery (at least 12 months prior to Day 1) or short-bowel
* syndrome.
* If taking probiotic supplements (enriched foods excluded), has been on a stable, well tolerated dose for at least 2 weeks prior to Day 1.
* Women of childbearing potential must have a negative pregnancy test (human chorionic
* gonadotropin) at screening and at baseline prior to the start of IMP.
* Screening laboratory evaluations (e.g., chemistry panel, complete blood count with
* differential, prothrombin time, urinalysis) and electrocardiogram (ECG) must be within
* normal limits or judged not to be clinically significant by the investigator. Subjects with
* known diabetes should be well controlled and have an A1c of ≤ 8% within 3 months prior to Day 1.
* Agree to abstain from tobacco/nicotine use for the duration of the inpatient stay.
* Subjects who are HIV positive, on therapy with normal CD4 counts and undetectable viral loads, can be included.

Exclusion Criteria:

* Acute or chronic medical (including COVID-19 infection), surgical, psychiatric, or social condition or laboratory abnormality (except those that can be explained by malabsorption) that may increase subject risk associated with study participation, compromise adherence to study procedures and requirements, or may confound interpretation of results and, in the judgment of the investigator, would make the subject inappropriate for enrollment.
* Estimated glomerular filtration rate < 45 mL/min/1.73 m2.
* History of kidney stones.
* Subjects taking supplements that contain vitamin C should continue to use their supplements at a constant dose throughout the study, having maintained a constant dose for 2 weeks prior to screening.
* Known primary hyperoxaluria.
* Pregnant or lactating.
* Administration or ingestion of any type of systemic (e.g., oral or intravenous) antibiotic within 5 half-lives of the agent prior to Day 1. Exception: topical antibiotics are allowed.
* Any co-morbid condition that may necessitate antibiotic use or disrupt the controlled diet during the study period.
* Intolerance of, or allergic reaction to, EcN, all PPIs, or any of the ingredients in SYNB8802v1 or placebo formulations.
* Dependence on alcohol or drugs of abuse.
* Current, immunodeficiency disorder including autoimmune, except for controlled HIV (see inclusion Criterion #9). disorders.
* Administration or ingestion of an investigational drug within 30 days or 5 half-lives, whichever is longer, prior to screening visit, or current enrollment in an investigational study.
* History of inflammatory bowel disease.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of SYNB8802v1, as assessed by measuring of vital signs | 17 days
  Vital Signs Resting vital signs will be collected as specified in the protocol. Subjects are required to remain in the sitting position for at least 5 minutes prior to obtaining vital signs. A symptom-directed physical examination will be performed by trained medical personnel as specified in the protocol.
Safety and tolerability of SYNB8802v1 by assessing clinical laboratory tests | 17 days
  The clinical laboratory tests listed in the protocol will be performed at the time points specified in the protocol's schedule of assessments.
Safety and tolerability of SYNB8802v1, as assessed by AEs, clinical laboratory tests, and vital sign measurements | 43 days
  Adverse events will be assessed continuously by direct observation and subject event recording and interviews. The severity of AEs will be evaluated using the NCI CTCAE, version 5.0 criteria.

SECONDARY OUTCOMES:
Change from baseline in 24-hour excreted UOx among SYNB8802v1-treated subjects versus those treated with placebo. | 17 days
  Urinary oxalate will be determined from 24-hour urine sample collections to be completed at the points specified in the Schedule of Assessments.

CONTACTS AND LOCATIONS:
Locations (1):
- PPD, part of Thermo Fisher Scientific, Austin, Texas, United States